CLINICAL TRIAL: NCT05100654
Title: Collaborative Urological Prosthetics Investigation Directive Research Group
Acronym: CUPID
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Loyola University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB19-1757
Record Dates: First submitted 2021-09-30; First posted 2021-10-29 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Erectile Dysfunction; Penile Prosthesis Infection
Keywords: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Doxycycline; Ciprofloxacin; Amoxicillin-Potassium Clavulanate Combination; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- No post-operative oral antibiotics (No Intervention): Patients will only receive 24hr of IV peri-operative antibiotics
- 6 days of oral antibiotics (Active Comparator): Patients will receive 24hr of IV peri-operative antibiotics and then 6 days of oral antibiotics
  Interventions: Drug: Doxycycline; Drug: Ciprofloxacin; Drug: Augmentin; Drug: Bactrim

INTERVENTIONS:
Drug: Doxycycline — Patients will be given 6 days of oral antibiotics based on local biograms, patient allergies and renal and liver function
  Arms: 6 days of oral antibiotics
Drug: Ciprofloxacin — Patients will be given 6 days of oral antibiotics based on local biograms, patient allergies and renal and liver function
  Arms: 6 days of oral antibiotics
Drug: Augmentin — Patients will be given 6 days of oral antibiotics based on local biograms, patient allergies and renal and liver function
  Arms: 6 days of oral antibiotics
Drug: Bactrim — Patients will be given 6 days of oral antibiotics based on local biograms, patient allergies and renal and liver function
  Arms: 6 days of oral antibiotics

SUMMARY:
The purpose of this study is to determine if an additional 6 days of oral antibiotics decreases the risk of penile prosthesis infection after implantation.

DETAILED DESCRIPTION:
Erectile dysfunction is a common problem and the incidence increases with age. Penile prosthesis placement for medication refractory erectile dysfunction is well established with high success rates. However, infection remains a dreaded complication with significant patient morbidity requiring device explant. Device innovations such as antibiotic coating and adaptations in technique have led to device infection rate reduction to ~1-3% in the hands of high volume implanters in modern series. The study team will perform a non-inferiority trial of post-operative antibiotic prophylaxis for IPP procedures with InhibiZonetm coated AMS 700 devices to confirm the hypothesis that a prolonged postoperative antibiotic regimen does not influence infection-related outcomes in de-novo IPP placement. The study team will determine potential risk factors for prosthetic infections and which patients would benefit from an extended post-operative oral antibiotic course of 6 days along with other objectives.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged 35 to 90 yo with no racial or ethnic restrictions and a diagnosis of erectile dysfunction.
2. Males clinically indicated for de-novo InhibiZonetm coated AMS 700 devices IPP placement procedure per local clinical guidelines who have elected to pursue penile prosthesis as an ED treatment.

Exclusion Criteria:

1. Patients with indwelling foreign body in the urinary tract > 24 hours prior to the procedure (i.e. foley catheter). Patients using clean intermittent catheterization will not be excluded.
2. Prior history of or current symptomatic urethral stricture.
3. History of cystitis caused by Tuberculosis.
4. Active Cytoxan/cyclophosphamide therapy or immunosuppressive systemic chemotherapy.
5. Prior augmentation cystoplasty or cystectomy.
6. Systemic neuromuscular disease known to affect the lower urinary tract such as Spinal Cord Injury, Multiple Sclerosis or other condition leading to neurogenic bladder.
7. Antibiotic use within the past 1 week or need for antibiotic management immediately prior to the study.
8. Cases where patients have had a prior penile prosthesis.
9. Any protected population (i.e. Prisoners)

Ages: 35 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Additional 6 days of oral antibiotics after Penile prothesis placement does not decrease the risk of device infection leading to surgical intervention | 12 months
  From day of surgery through 1 year we are hoping to show that additional 6 days of oral antibiotics do not decrease the risk of penile prosthesis infection requiring surgical intervention for device removal.

SECONDARY OUTCOMES:
Additional 6 days of oral antibiotics after Penile prosthesis placement does not decrease the risk of superficial tissue infections after penile prothesis implantation. | 12 months
  From day of surgery through 1 year we are hoping to show that additional 6 days of oral antibiotics do not decrease the risk of superficial skin infection after penile prosthesis placement.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Faris, MD, Principal Investigator — University of Chicago Department of Surgery
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share individual participant data that is de-identified available to all qualified investigators
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Upon publication of the major manuscript to be generated from this study. Data will be deposited in an appropriate major database
Access Criteria: All qualified investigators who sign appropriate data use agreements with the University of Chicago